CLINICAL TRIAL: NCT02977858
Title: Interactive Spaced Education Game to Support Constipation Management in Pediatric Primary Care
Brief Title: ISE to Support Constipation Management
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-9317
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2018-07

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dissemination: Educational practice for HCPs,Dissemination only - Practices who will participate in education for constipation management guidelines via dissemination of webinar alone.
  Interventions: Other: Educational practice for HCPs,Dissemination only
- Dissemination + ISE: Educational practice for HCPs,Spaced Education - Practices who will participate in education for constipation management guidelines via dissemination of webinar along with a web-based format referred to as Interactive Spaced Education.
  Interventions: Other: Educational practice for HCPs,Dissemination only; Other: Educational practice for HCPs,Spaced Education

INTERVENTIONS:
Other: Educational practice for HCPs,Dissemination only — Study participants are health care professionals (HCPs) who will be provided educational material and complete knowledge assessments
Other: Educational practice for HCPs,Spaced Education — Study participants are health care professionals (HCPs) who will be provided educational material via a Spaced Education program; participants will subsequently complete knowledge assessments
  Groups: Dissemination + ISE

SUMMARY:
This study is a single site prospective controlled trial assessing two educational interventions designed to educate local pediatric Primary Care Physicians (PCP) and nurses on collaboratively developed treatment guidelines for pediatric constipation. The study aims to assess the impact of an Spaced Education game to aid the implementation of the management guideline. PCP adherence to recommended treatment will be assessed in addition to PCP satisfaction with the educational methods, constipation knowledge and patient outcomes.

DETAILED DESCRIPTION:
Primary care practices in the Greater Cincinnati region, that are part of the Ohio Valley Pediatric Care Association (OVPCA) will be recruited to take part in the study. It is estimated that approximately 170 providers in 40 practices will take part overall. The study participants will be the PCPs and nurses in their practices.

Prior to the educational intervention (described below), participating PCPs and nurses will be asked to complete Constipation Action Plan (CAP) forms detailing the treatments they prescribed to each patient with constipation symptoms at each new visit and the subsequent follow up visits for constipation. The CAP form will contain a section to describe the patient's symptoms as well as fields to be checked for each treatment the PCP instructed the patient to follow.

Practices will be clustered by size (number of providers) and randomly assigned to 1 of 2 educational interventions (Dissemination or Dissemination +Interactive Spaced Education).

Dissemination will include webinars and e-mail distribution of the Constipation Management Guideline and a slide set containing the evidence-based rationale as well as clinical tips for advanced management of functional constipation. All PCPs will receive the guideline and slide set and be offered an opportunity to ask questions of a gastroenterologist.

Participating PCPs and nurses randomized to the Interactive Spaced Education (ISE) arm will complete an online ISE course assessing their understanding of the constipation guidelines.

Constipation knowledge will be tested via quiz in multiple choice format. Online surveys to assess satisfaction with the educational intervention, likelihood to change practice, ease of participation in the SE course (if applicable) and feedback for ways to improve future educational efforts will be administered at three time-points.

ELIGIBILITY:
Inclusion Criteria:

* PCPs and nurses who are willing and able to complete the education intervention throughout the study time-frame, as outlined in the protocol (education intervention does not need to be completed prior to taking part in the study)
* PCPs and nurses who are willing to complete Constipation Action Plans and submit them in a timely fashion to the CCHMC Quality Improvement program staff

Exclusion Criteria:

* PCPs or nurses who are unwilling and/or unable to follow protocol requirements.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care practices in the Greater Cincinnati region, that are part of the Ohio Valley Pediatric Care Association (OVPCA) will be recruited to take part in the study. It is estimated that approximately 170 providers in 40 practices will take part overall. The study participants will be the PCPs and nurses in their practices
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Patient Referral | 2 years
  Determine if online ISE reduces referrals of patients with constipation to pediatric gastroenterologists

SECONDARY OUTCOMES:
Improved knowledge gains | 2 years
  Determine if online ISE in addition to dissemination improves knowledge gains by pediatricians and medical staff
Improved adherence to Constipation Management Guideline | 2 years
  Determine if online ISE in addition to dissemination improves adherence by pediatricians to the Constipation Management Guideline

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mallon, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mallon D, Fei L, Farrell M, Anderson JB, Klein M. Randomized Controlled Trial of Interactive Spaced Education to Support Constipation Management by Pediatric Primary Care Providers. J Pediatr Gastroenterol Nutr. 2022 May 1;74(5):568-574. doi: 10.1097/MPG.0000000000003405. PMID 35149642